CLINICAL TRIAL: NCT06723106
Title: Phase 1b Open-label, Long-term Extension Basket Trial of RAY121 to Inhibit Classical Complement Pathway in Immunological Diseases (RAINBOW-LTE Trial)
Brief Title: Phase 1b Long-term Extension Trial of RAY121 in Immunological Diseases (RAINBOW-LTE Trial)
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAY903CT
Record Dates: First submitted 2024-11-27; First posted 2024-12-09 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Antiphospholipid Syndrome (APS); Bullous Pemphigoid (BP); Behçet's Syndrome (BS); Dermatomyositis (DM); Immune-mediated Necrotizing Myopathy (IMNM); Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Antiphospholipid Syndrome; Pemphigoid, Bullous; Behcet Syndrome; Dermatomyositis; Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RAY121 (Experimental): All enrolled patients will receive RAY121 multiple dose
  Interventions: Drug: RAY121

INTERVENTIONS:
Drug: RAY121 — Injection

SUMMARY:
This is a long-term extension trial of RAY121 in patients with immunological diseases such as antiphospholipid syndrome (APS), bullous pemphigoid (BP), Behçet's Syndrome (BS), dermatomyositis (DM), immune-mediated necrotizing myopathy (IMNM) and immune thrombocytopenia (ITP).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Have completed 4 doses of RAY121 administrations in RAY902CT trial and shown clinical responses
3. Ability to comply with the study protocol, in the investigator's judgment
4. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use highly effective contraceptive methods during the treatment period and 20 weeks (140 days) after the last dose of RAY121
5. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

1. History of anaphylaxis or hypersensitivity to a biologic agent
2. Known active infection with encapsuled bacteria
3. History of Neisseria meningitidis infection
4. Planned surgery
5. Pregnant or breastfeeding, or intending to become pregnant
6. Clinically significant electrocardiogram abnormalities
7. Illicit drug or alcohol abuse
8. Known or suspected immune deficiency
9. Treatment with investigational therapy other than RAY121
10. Vaccination with a live vaccine within 4 weeks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Baseline to Week 52
  Incidence, severity, and causal relationship of AEs

SECONDARY OUTCOMES:
RAY121 concentration | Baseline to Week 52
  Serum RAY121 concentration
Change from baseline in active C1s | Baseline to Week 52
  Concentration of active C1s will be measured and assessed against baseline values
Change from baseline in total C1s | Baseline to Week 52
  Concentration of total C1s will be measured and assessed against baseline values
Change from baseline in complement activity (classical pathway) | Baseline to Week 52
  Level of complement activity (classical pathway) will be measured and assessed against baseline values
Anti-RAY121 antibodies | Baseline to Week 52
  Titer of anti-RAY121 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co.Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (54):
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Campbelltown Public Hospital, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - Box Hill Hospital, Melbourne, Victoria
- AKH - Medizinische Universitaet Wien, Abteilung fuer Klinische Pharmakologie, Vienna, Austria
- Bulgaria (3):
  - Diagnostic Consultation Center CONVEX EOOD, Sofia, Sofia City Province
  - "SHATHD" EAD Sofia, Sofia, Sofia City Province
  - UMHAT "Prof. Dr. St. Kirkovich", AD, Stara Zagora, Stara Zagora Province
- DiIEX Recherche Sherbrooke, Inc, Sherbrooke, Quebec, Canada
- Croatia (3):
  - Clinical Hospital Center "Sestre Milosrdnice", Zagreb, City of Zagreb
  - University hospital centre Zagreb, Zagreb, City of Zagreb
  - Specialty Hospital Medico, Rijeka, Primorje-Gorski Kotar County
- Sanatorium Profesora Arenbergera, Prague, Prague, Czechia
- France (2):
  - Hopital Lapeyronie,Service d'Immuno Rhumatologie, Montpellier, Occitanie
  - AP-HP Hôpital Universitaire Pitié Salpêtrière, Paris, Île-de-France Region
- Germany (5):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Klinik und Poliklinik f. Dermatologie, Sachsen, Bundesländer
  - Universitaetsmedizin Goettingen, Göttingen, Göttingen District
  - Universitaetsklinikum Schleswig Holstein - Campus Luebeck, Klinik f Dermatologie, Allergologie u Venerologie, Lübeck, Schleswig-Holstein
- Hungary (2):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged, Csongrád-Csanád County
  - Semmelweis Egyetem, Budapest
- Italy (3):
  - IRCCS Istituto Scientifico Romagnolo Per Lo Studio Dei Tumori "Dino Amadori" - IRST, Meldola, Forlì-Cesena Province
  - Istituto Clinico Humanitas, Milan, Milan Province
  - Ospedale San Giovanni Bosco, Torino, Turin Province
- Japan (8):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tohoku University Hospital, Sendai, Miyagi
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - Okayama University Hospital, Okayama
- Netherlands (2):
  - University Medical Centre Groningen UMCG, Groningen, Groningen Province
  - UMC Utrecht, Utrecht, Utrecht Province
- Norway (2):
  - Sorlandet sykehus Kristiansand, Kristiansand, Agder County
  - Stavanger Universitetssjukehus, Stavanger, Rogaland County
- Institute Reumatologii I'm. Eleonory Reicher, Warsaw, Masovian Voivodeship, Poland
- Portugal (2):
  - Centro Clinico Academico Braga, Braga, Braga District
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E., Vila Nova de Gaia, Porto District
- Romania (2):
  - Centrul Medical Monza SRL, Bucharest, Bucharest Municipality
  - Oncology Institute Prof. Dr. Ion Chiricuta I.O.C.N., Cluj-Napoca, Cluj
- Spain (7):
  - Clinica Universidad de Navarra, Pamplona, Community of Madrid & Navarre
  - Hospital Universitario Ramon y Cajal, Servicio de Reumatologia, Madrid, Madrid
  - Hospital Universitario 12 de October, Madrid, Madrid
  - Hospital Universitari Vall d'Hebron, Internal Medicine Dept., Barcelona, Province of Barcelona and Catalonia
  - Hospital Universitario Reina Sofia, Córdoba, Province Of Córdoba
  - Hospital Universitario Virgen del Rocio, Seville, Province Of Seville
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taichung Veterans General Hospital, Taipei
- Turkey (Türkiye) (2):
  - Dr. Abdurrahman Yurtaslan Oncology Teaching and Research Hospital, Ankara, Ankara
  - Istanbul University Istanbul Medical Faculty, Istanbul, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform. For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).